CLINICAL TRIAL: NCT04933448
Title: Ketogenic Diet Following Moderate to Severe Pediatric Traumatic Brain Injury: A Pilot Study
Brief Title: Ketogenic Diet Following Moderate to Severe Pediatric Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gillette Children's Specialty Healthcare (Other)
Collaborators: State of Minnesota Spinal Cord Injury and Traumatic Brain Injury Research Grant Program (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009115
Record Dates: First submitted 2021-06-17; First posted 2021-06-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prospective Intervention Group (Experimental): Participants will receive standard of care for acute management of moderate to severe traumatic brain injury, together with a weight-based ketogenic diet added for up to fourteen days.
  Interventions: Other: Ketogenic Diet
- Historical Control Group (No Intervention): Medical records of past TBI patients will be used as controls matched for age, gender, socioeconomic status (type of health care coverage including private insurance vs. government-funded coverage), lowest first 24 hour post-injury Glasgow Coma Score (GCS) (<8 or 8-12), and pre-injury school program (regular or special education).

INTERVENTIONS:
Other: Ketogenic Diet — The ketogenic diet (KD) is an alternative feeding regimen that has been in use since 1921. It is a high-fat, low carbohydrate, and moderate protein diet. There are various forms of the KD. The classic KD consists of long-chain triglycerides with a fat-to-combined-protein-and-carbohydrate ratio that can vary. At the investigating institution, it is standard of care to initiate a ketogenic diet at a ratio of 2:1, and to increase the ratio to 3:1 or 4:1 as needed to achieve ketosis.
  Other Names: Keto
  Arms: Prospective Intervention Group

SUMMARY:
The primary objective of this study is to evaluate the feasibility and safety of using the ketogenic diet (KD) in children who sustained moderate to severe traumatic brain injury (TBI). The secondary objective is a preliminary evaluation of the outcomes of children who have had the standard of care plus the KD, compared to those with standard of care alone. Outcome measures for the secondary objective will include: need for ventriculoperitoneal shunt, duration of unconsciousness, need for any type of craniotomy, duration of post-traumatic amnesia, acute hospitalization length of stay, and cognitive and motor function at 12 months after injury. If this study demonstrates feasibility and safety, the information related to outcomes will be used to inform the planning of a future, larger, randomized study of the efficacy of the KD in children and adolescents with TBI. Specifically, this information will be used to assist with sample size calculations for this future study.

DETAILED DESCRIPTION:
The KD is an alternative feeding regimen that has been in use since 1921. It is a high fat, low carbohydrate and moderate protein diet. There are various forms of the KD. The classic KD consists of long-chain triglycerides with a fat-to-combined-protein-and-carbohydrate ratio that can vary. At our institution, it is standard of care to initiate a ketogenic diet at a ratio of 2:1, and to increase the ratio to 3:1 or 4:1 as needed to achieve ketosis. Clinically, the KD has been proven to be an effective therapy in children and adolescents with refractory epilepsy, as well as for those with type II diabetes. In addition, an international consensus was published in 2009 that recommended the use of the KD to treat epilepsy refractory as an alternative to at least two antiepileptic medications. Before initiating the KD for epilepsy management, labs such as urine and blood ketones, blood glucose and a basic metabolic panel including magnesium are commonly recommended. Risks for long-term use of the KD include but are not limited to the following: hypercholesterolemia, mineral deficiencies, acidosis, constipation, weight loss and nephrolithiasis. However, short-term use should significantly limit the occurrence of these potential complications.

ELIGIBILITY:
Inclusion Criteria:

* Age limits met at the time of injury and admission
* Participants with moderate to severe traumatic brain injury defined as a Glasgow Coma Scale Score of 3-12 (lowest score in the first 24 hours after injury). Individuals requiring craniotomy and/or evacuation of intracranial hemorrhage may be included.

Exclusion Criteria:

* Currently on an oral diet at time of screening or currently on IV-only and in opinion of Pediatric Intensive Care Unit intensivist will be transitioning to an oral diet, not tube-feeding
* Anoxia/ischemia as a significant portion of injury, including near-drowning
* Non-accidental traumatic brain injury (i.e., assault, abuse)
* Penetrating injury including gunshot wounds
* Pregnancy
* Any condition that in the opinion of the Pediatric Intensive Care Unit or neurosurgery medical staff warrants exclusion from the study

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Ability to complete a course of the ketogenic diet (KD) | 14 days
  Safety and feasibility will be determined by the ability to complete a 14-day course of the KD after TBI without needing to terminate the diet due to intolerance resulting from gastrointestinal side effects (for example, nausea and vomiting, diarrhea, or acidosis), or due to abnormal findings on laboratory tests. Outcome is reported as the number of participants who complete the 14-day keto diet treatment.

SECONDARY OUTCOMES:
Duration of Unconsciousness | 14 days
  Outcome is reported as the length of time (in hours) a participant is unconscious following their injury.
Need for Surgeries | 14 days
  Outcome is reported as the number of surgeries required in each group following injury.
Duration of Acute Hospitalization | 14 days
  Outcome is reported as the length (in days) of acute hospitalization following injury.
Duration of Post-traumatic Amnesia | 14 days
  Outcome is reported as the length of time (in days) that a participant experiences amnesia following their injury.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Krach, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation; Angela Sinner, DO, Principal Investigator — Department of Physical Medicine and Rehabilitation
Locations (2):
- United States (2):
  - Children's Minnesota, Minneapolis, Minnesota
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
pilot, feasibility study only.